CLINICAL TRIAL: NCT06979973
Title: A Phase 1, Open-label, Drug-Drug Interaction Study to Assess the Pharmacokinetic Interactions Between CKD-508, Midazolam, and Rosuvastatin in Healthy Adult Male Participants
Brief Title: A Drug-drug Interaction Study to Investigate the Pharmacokinetic Interactions Between CKD-508, Midazolam, and Rosuvastatin in Healthy Adult Male Participants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A104_03DDI2501
Record Dates: First submitted 2025-05-09; First posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam, Rosuvastatin, CKD-508 (Experimental): Single dose of Midazolam Single and Multiple dose of Rosuvastatin Multiple dose of CKD-508
  Interventions: Drug: Midazolam; Drug: Rosuvastatin; Drug: CKD-508 Tablet

INTERVENTIONS:
Drug: Midazolam — midazolam syrup
Drug: Rosuvastatin — Rosuvastatin
Drug: CKD-508 Tablet — CKD-508

SUMMARY:
Phase 1, open-label, non-randomized, three-treatment, one-sequence interaction study to evaluate the PK interactions between CKD-508, midazolam, and rosuvastatin in healthy adult male participants

ELIGIBILITY:
Inclusion Criteria:

* The participant is capable of providing signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and the protocol.
* Male adults aged 18 to 45 years at screening.
* Healthy participants were determined by pre-study medical evaluation and judged by the Investigator.
* Non-smoker (or other nicotine use) as determined by history (no nicotine use over the past 6 months) and by urine cotinine concentration (<200 ng/mL) at screening and admission.

Exclusion Criteria:

* History or evidence of clinically significant cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder as determined by the Investigator.
* Presence of any disorder that would interfere with the absorption, distribution, metabolism, or excretion of study intervention as judged by the Investigator.
* Serum alkaline phosphatase (ALP) or total bilirubin ≥upper limit of normal (ULN), or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >ULN at either screening or admission.
* Abnormal renal function with estimated glomerular filtration rate (eGFR) <80 mL/min/1.73 m2 at screening.
* History or presence of clinically significant abnormal cardiac automaticity, heart rhythm, ECG findings, or other relevant conditions that may pose a risk to the participants as judged by the Investigator.
* Resting heart rate ≥100 bpm or <50 bpm at screening or admission.
* Resting systolic blood pressure ≥140 mmHg and /or diastolic blood pressure ≥90 mmHg at screening or admission.
* Evidence of known risk factors for atrial fibrillation (eg, smoking, hyperthyroidism, diabetes)
* History of alcohol and/or illicit drug abuse within 2 years before screening or positive urine test for alcohol or positive urine drug test at screening or admission.
* Positive test for HBsAg, HCV RNA, or HIV antibody at screening.
* Donation of blood (>500 mL) or blood products within 2 months prior to dosing.
* Use of over-the-counter medications (including vitamins), prescription medications, or herbal remedies within 14 days or 5 half-lives, whichever is longer, prior to dosing.
* Receiving an investigational drug within 30 days or >5 half-lives of the investigational drug, whichever is longer, prior to dosing.
* History of hypersensitivity to CETP inhibitor or statins or midazolam or to medicinal products with similar chemical structures.
* Individual unlikely to comply with the protocol requirements, instructions, and study-related restrictions.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-14 (Estimated); Primary Completion 2025-08-16 (Estimated); Study Completion 2025-08-16 (Estimated)

PRIMARY OUTCOMES:
Cmax of midazolam | 24 hours
  Maximum plasma concentrations of midazolam after single dose
AUClast of midazolam | 24 hours
  Area under the concentration-time curve of midazolam after single dose
AUCinf of midazolam | From 0 hours to 24 hours on Day 1 and Day 24
  Area under the concentration-time curve extrapolated to infinity of midazolam
Cmax of Rosuvastatin | 72 hours
  Maximum plasma concentrations of rosuvastatin after single dose
AUClast of rosuvastatin | 72 hours
  Area under the concentration-time curve of rosuvastatin after single dose
AUCinf of rosuvastatin | From 0 hours to 72 hours on Day 1 and Day 24
  Area under the concentration-time curve extrapolated to infinity of rosuvastatin
Cmax,ss of CKD-508 | 24 hours
  Maximum plasma concentration at steady state of CKD-508
AUCtau,ss of CKD-508 | 24 hours
  Area under the concentration time curve until the end of dosing interval at steady state of CKD-508
Cmin,ss of CKD-508 | 24 hours
  Minimum plasma concentration at steady state of CKD-508

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Glendale, California, United States